CLINICAL TRIAL: NCT05729308
Title: Comparative Study Between Caudal Epidural Block and Bilateral Erector Spinae Plane Block in Adult Patients Undergoing Lumbosacral Spine Surgeries.
Brief Title: Comparative Study Between Caudal Epidural Block and Bilateral Erector Spinae Plane Block in Lumbosacral Spine Surgeries.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: md 335/2022
Record Dates: First submitted 2023-01-28; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (CE): Patients receiving caudal epidural block (Active Comparator)
  Interventions: Procedure: caudal epidural block
- Group (ESP): Patients receiving bilateral erector spinae plane block. (Active Comparator)
  Interventions: Procedure: bilateral erector spinae plane block
- Group (C): Control group, patients receiving general anesthesia with intravenous analgesia. (Active Comparator)
  Interventions: Procedure: general anesthesia with intravenous analgesia.

INTERVENTIONS:
Procedure: caudal epidural block — The patient will be positioned in prone position, sterilized from the iliac crest margin to the lower buttock. Sacral horns will be palpated and sacral hiatus and epidural area will be determined at S4-S5 level through the ultrasound guidance using SonoSite M Turbo(USA).The scanning probe is the linear multi-frequency 6-13 MHz transducer (L25 x 6-13 megahertz linear array)that is covered in sterile plastic bag.Short axis (transverse view) is used first to identify the two sacral cornua as two hyperechoic reverse U-shaped structure "Frog sign" and the sacrococcygeal ligament in between and epidural space beneath. An 18-gauge epidural needle (length 90 mm) is used for direct puncture of sacrococcygeal membrane out of plane then the probe is rotated to long axis (longitudinal view) and the needle is seen in plane in the epidural space. Injection of 30 ml 0.25% bupivacaine will expand the epidural space
  Arms: Group (CE): Patients receiving caudal epidural block
Procedure: bilateral erector spinae plane block — The patient will be in the prone position, after skin sterilization, ESP block will be performed at the level of T12. A curvilinear high-frequency ultrasound transducer will be placed sagittal 3 cm lateral to T12 spinous process where a hyperechoic shadow of the transverse process (TP) and erector spinae will be defined. A 22-gauge spinal needle will be inserted in cranial to caudal direction toward TP in plane to the ultrasound transducer until the needle touches the TP crossing the whole muscles. The location of the needle tip will be confirmed by visible normal saline solution separating erector spinae muscle off the bony shadow of the TP on ultrasound imaging. After confirming the needle site, 15 mL of 0.25% bupivacaine will be injected. The procedure will be repeated following the same steps on the other side
  Arms: Group (ESP): Patients receiving bilateral erector spinae plane block.
Procedure: general anesthesia with intravenous analgesia. — * Multimodal therapy with acetaminophen, and nonsteroidal anti-inflammatory drugs (NSAIDs) will be used.
  * Vital data will be monitored as mentioned Intraoperatively, if the pulse rate and/or mean blood pressure increased above 20% of the baseline, IV fentanyl will be administered as an incremental dose of 50 µg.
  * The patients will be monitored for heart rate and blood pressure at regular 10-minute intervals. If blood pressure decreased more than 20% from baseline, then the patient will receive 500 mL saline infusion; if no response is seen, then 5 mg ephedrine will be administered. If heart rate decreased to 45 beats per minute, an IV injection of 0.1 mg /kg atropine will be administered.
  Arms: Group (C): Control group, patients receiving general anesthesia with intravenous analgesia.

SUMMARY:
It is widely believed that major lumbosacral spine surgeries are associated with severe postoperative pain that may delay the functional recovery of the patient. Caudal epidural injection (CE) has an important role in providing effective pain relief post lumbosacral spine surgeries by blocking sensory input at the level of the spinal cord. Erector Spinae Plane Block (ESPB) is a relatively new technique of trunk fascial block which was introduced in 2016. Reports showed that ESPB significantly relieved postoperative pain in patients with lumbosacral spine surgery, reducing the use of analgesics.The overall benefit of intravenous (IV) analgesia versus pre-emptive analgesia by caudal epidural or erector spinae block is still controversial.

The aim of this study is to compare the pre-emptive analgesic effect of bilateral erector spinae plane block versus Caudal epidural analgesia versus the conventional intravenous analgesia in adult patients undergoing lumbosacral spine surgeries under general anesthesia.

DETAILED DESCRIPTION:
78 Participants undergoing lumbosacral spine surgeries who met the inclusion criteria will be divided into three groups each group contains 26 patients:

Group (CE): Patients receiving caudal epidural block. Group (ESP): Patients receiving bilateral erector spinae plane block. Group (C): Control group, patients receiving general anesthesia with intravenous analgesia.

• Study procedures:

* Routine preoperative assessment will be done for all the participants.
* All participants will be fasting before the procedure not less than 6 hours.
* General anesthesia will be induced with midazolam (0.05mg/kg), propofol (1.5-2mg/kg), fentanyl (1-2μg/kg) and atracurium (0.5mg/kg),
* Tracheal intubation will be performed. After induction, general anesthesia will be maintained with a volatile anesthetic agent (0.9:1.2% isoflurane) and controlled ventilation with atracurium every 20 mins (0.1 mg/kg).
* Standard monitoring of mean arterial blood pressure (MAP), heart rate (HR) and peripheral pulse oximeter (SPO2) value will be monitored at time of induction (time 0) and every 10 minutes till the end of the procedure.

Group (CE): Caudal epidural group The patient will be positioned in prone position, sterilized from the iliac crest margin to the lower buttock. Sacral horns will be palpated and sacral hiatus and epidural area will be determined at S4-S5 level through the ultrasound guidance using SonoSite M Turbo(USA).The scanning probe is the linear multi-frequency 6-13 megahertz transducer (L25 x 6-13 megahertz linear array)that is covered in sterile plastic bag.Short axis (transverse view) is used first to identify the two sacral cornua as two hyperechoic reverse U-shaped structure "Frog sign" and the sacrococcygeal ligament in between and epidural space beneath. An 18-gauge epidural needle (length 90 mm) is used for direct puncture of sacrococcygeal membrane out of plane then the probe is rotated to long axis (longitudinal view) and the needle is seen in plane in the epidural space. Injection of 30 ml 0.25% bupivacaine will expand the epidural space.

Group (ES): Erector spinae group The patient will be in the prone position, after skin sterilization, ESP block will be performed at the level of T12. A curvilinear high-frequency ultrasound transducer will be placed sagittal 3 cm lateral to T12 spinous process where a hyperechoic shadow of the transverse process (TP) and erector spinae will be defined. A 22-gauge spinal needle will be inserted in cranial to caudal direction toward TP in plane to the ultrasound transducer until the needle touches the TP crossing the whole muscles. The location of the needle tip will be confirmed by visible normal saline solution separating erector spinae muscle off the bony shadow of the TP on ultrasound imaging. After confirming the needle site, 15 mL of 0.25% bupivacaine will be injected. The procedure will be repeated following the same steps on the other side.

Group(C): General anesthesia with conventional intravenous analgesia.

* Multimodal therapy with acetaminophen, and nonsteroidal anti-inflammatory drugs (NSAIDs) will be used.
* Vital data will be monitored as mentioned Intraoperatively, if the pulse rate and/or mean blood pressure increased above 20% of the baseline, IV fentanyl will be administered as an incremental dose of 50 µg.
* The patients will be monitored for heart rate and blood pressure at regular 10-minute intervals. If blood pressure decreased more than 20% from baseline, then the patient will receive 500 mL saline infusion; if no response is seen, then 5 mg ephedrine will be administered. If heart rate decreased to 45 beats per minute, an IV injection of 0.1 mg /kg atropine will be administered.
* After completion of the surgical procedure, patient will be in supine position, isoflurane will be discontinued and fresh gas flow will be increased and any residual neuromuscular blockade will be reversed by I.V neostigmine 50 μg/kg (to a maximum of 5 mg) plus atropine 10-20 μg/kg.
* Any blood and secretions in the pharynx will be carefully suctioned. Tracheal extubation will be performed when the patient regained consciousness, has sufficient spontaneous breathing, intact gag reflex, purposeful movement, and spontaneous eye opening.
* After extubation in the three groups, the patients will be transferred to the postanesthesia care unit and will be monitored as mentioned above.
* The visual analog score (VAS) is a validated, subjective measure for acute pain. Scores are recorded by making a handwritten mark on a 10 cm line that represents a continuum between "no pain" and "worst pain".
* VAS score will be assessed at 15 & 30 mins, then at 2, 6, 12, 24 hours post-operatively.
* Rescue pain analgesia will be given postoperatively for visual analogue scale (VAS)≥4 by nalbuphine hydrochloride (Nalufin)10-20 mg/70kg IV q3-6hr on demand; individual dose not to exceed 20 mg). VAS will be reassessed 15 minutes later to any post analgesic injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for lumbosacral spine surgery level from L4 to S1.
* American Society of Anesthesiologists classification (ASA) class I or II.

Exclusion Criteria:

* Refusal of procedure or participation in the study.
* American Society of Anesthesiologists classification (ASA) class III or IV.
* Coagulation disorders (platelets count < 100,000; International normalized ratio >1.4; Patient control time< 60%) and coagulopathies.
* Skin lesion or infection at the injection site.
* Known allergy to any of the medications used.
* Chronic opioid users.
* Patients with pre-operative opioid consumption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
postoperative analgesia | immediately postoperative
  using the visual analogue scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
postoperative analgesia | 2 hours postoperative
  using the visual analogue scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
postoperative analgesia | 6 hours postoperative
  using the visual analogue scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
postoperative analgesia | 12 hours postoperative
  using the visual analogue scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
postoperative analgesia | 24 hours postoperative
  using the visual analogue scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')

SECONDARY OUTCOMES:
intraoperative mean arterial blood pressure | every 10 minutes intraoperative till end of surgery
  measured by non invasive blood pressure monitoring
intraoperative heart rate | every 10 minutes intraoperative till end of surgery
  measured by twelve leads electrocardiogram
postoperative first rescue analgesia time | during the 24 hours postoperative
Surgical field bleeding. | from the start till the end of the operation
  using Fromme score assessed by the surgeon 6-point scale
  Endoscopic surgical field grading system
  Grade Assessment 0 No bleeding (cadaveric conditions)
  1. Slight bleeding, no suctioning required
  2. Slight bleeding, occasional suctioning required
  3. Slight bleeding, frequent suctioning required; bleeding threatens surgical field a few seconds after suction is removed
  4. Moderate bleeding, frequent suctioning required, and bleeding threatens surgical field directly after suction is removed
  5. Severe bleeding, constant suctioning required; bleeding appears faster than can be removed by suction; surgical field severely threatened and surgery usually not possible
Number of participant with postoperative nausea | during the 24 hours postoperative
Number of participant with postoperative vomiting | during the 24 hours postoperative
Number of participant with postoperative urinary retention | during the 24 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No